CLINICAL TRIAL: NCT00821626
Title: Utility of Rapid Flu Tests in the Medical Management of Returning Travelers With Fever
Brief Title: Rapid Flu Tests in Travelers With Fever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Serge de Valliere, Consultant, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PMU-Flu
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Influenza
Keywords: Influenza; Rapid flu test; Returning travelers with fever
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid test (Active Comparator): Returning travelers with fever will have a rapid flu test
  Interventions: Device: BD Directigen EZ Flu A+B
- Comparator (Sham Comparator): Returning travelers with fever will benefit of the usual medical care, without rapid flu test
  Interventions: Other: Control

INTERVENTIONS:
Device: BD Directigen EZ Flu A+B — Naso-pharyngeal swab and rapid flu test
  Other Names: BD Directigen EZ Flu A+B, serial number 8010589
  Arms: Rapid test
Other: Control — No rapid flu test
  Arms: Comparator

SUMMARY:
Influenza is a frequent cause of fever in returning travelers. Usually diagnosis rests on the clinical picture. Rapid flu tests are becoming increasingly popular, although their sensitivity and specificity are suboptimal. The objective of this study is to evaluate if rapid flu tests influence the medical management of returning travelers with fever, a population at intermediate risk for influenza infections.

DETAILED DESCRIPTION:
Travelers are at risk of acquiring infectious diseases. Previous studies have estimated that about 11% of travelers develop fever during or shortly after their trip abroad. Influenza has been shown to be one of the most important cause of fever amongst travelers. A sero-epidemiological survey showed that 27 of 211 patients (12.8%) with fever during or after a trip abroad developed antibodies against the influenza virus. Another study showed that 13% of travellers, who consulted after return with flu-like symptoms, had PCR or culture-proven influenza. The incidence of influenza in travellers varies according to the seasons, but cases can be seen year round. In tropical countries transmission is year-long and in the southern hemisphere the flu epidemics occur during the summer of the northern hemisphere.

In most hospitals no confirmatory test for influenza is routinely done. For special cases a PCR or viral culture can be requested, but the results are only available after 48 hours for the PCR and after several days for the culture. It is suspected that the inability to confirm the diagnosis of flu contributes to the request of a greater number of useless investigations and inappropriate use of anti-infective treatments.

Rapid diagnostic tests are easy to use, relatively cheap and they yield a result within a clinically relevant time frame (30 minutes). For the detection of influenza there are a variety of rapid diagnostic tests on the market. The reported sensitivities and specificities are quite variable, but the new generations report median sensitivities of 70 - 75% and median specificities between 90 and 95%. The rapid tests are considered most useful in patient populations with a significant proportion of influenza cases. The WHO encourages to use rapid diagnostic tests for influenza in returning travelers with fever, considering that this patient population is at significant risk of acquiring influenza during their trip.

The aim of this study is to evaluate if rapid flu tests influence the medical management of returning travelers with fever

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Returning from abroad within the last 14 days
* Documented fever of 38oC or above or anamnestic fever + cough or sore throat within the last 4 days before the consultation.

Exclusion Criteria:

* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serge de Valliere, MD, Principal Investigator — Medical Outpatient Clinic, University Hospital of Lausanne
Locations (2):
- Switzerland (2):
  - Tropical Institute Basel, Basel
  - Medical outpatient clinic, University Hospital of Lausanne, Lausanne

REFERENCES:
- [Derived] Berthod D, Genton B, Hatz C, Blum J, de Valliere S. Ability of physicians to diagnose influenza and usefulness of a rapid influenza antigen test in febrile returning travelers: A randomized controlled trial. Travel Med Infect Dis. 2015 Sep-Oct;13(5):394-9. doi: 10.1016/j.tmaid.2015.08.001. Epub 2015 Aug 28. PMID 26358968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between January 2009 and November 2012.
Groups:
- Rapid Test: Returning travelers with fever will have a rapid flu test BD Directigen EZ Flu A+B done on a a naso-pharyngeal swab
Period: Overall Study
Arm/Group | Rapid Test | Comparator
Started | 60 | 33
Completed | 60 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rapid Test: Returning travelers with fever will have a rapid flu test BD Directigen EZ Flu A+B done on a naso-pharyngeal swab
- Total: Total of all reporting groups
Arm/Group | Rapid Test | Comparator | Total
Number analyzed (Participants) | 60 | 33 | 93
Age, Continuous [Median (Full Range); unit: years] | 35 [18 to 79] | 35 [18 to 70] | 35 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 15 | 43
  Male | 32 | 18 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 60 | 33 | 93

OUTCOME MEASURES:

1. Primary Outcome: Cost for the Medical Management of Patients
Time Frame: 4 years
Measure: Mean (95% Confidence Interval); unit: USD
Groups:
- Rapid Test: Returning travelers with fever will have a rapid flu test (BD Directigen EZ Flu A+B) on a naso-pharyngeal swab
Arm/Group | Rapid Test | Comparator
Number analyzed (Participants) | 60 | 33
USD | 581 [454 to 707] | 661 [522 to 800]

2. Secondary Outcome: Chest X-ray Requested
Description: Number of patients for whom a chest X-ray was requested as part of the medical management
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Test | Comparator
Number analyzed (Participants) | 60 | 33
Participants | 9 | 2

3. Secondary Outcome: Number of Patients Receiving a Prescription for Antibiotics
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Test | Comparator
Number analyzed (Participants) | 60 | 33
Participants | 14 | 13

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Rapid Test | Comparator
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/33
Other Adverse Events (participants affected / at risk) | 0/60 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No